CLINICAL TRIAL: NCT04948684
Title: Efficacy of Botulinum Toxin for the Treatment of Dystonia Associated With Parkinson's Disease and Atypical Parkinsonism: a Monocentric Cohort Study With Patient Reported Outcome
Brief Title: Efficacy of Botulinum Toxin for the Treatment of Dystonia Associated With Parkinson's Disease and Atypical Parkinsonism
Status: Completed | Type: Observational
Sponsor: Hospital Avicenne (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Principal Investigator, Arnaud Lapostolle, interne, Hospital Avicenne
Other Study IDs: CLEA-2021-167
Record Dates: First submitted 2021-06-06; First posted 2021-07-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Parkinson Disease; Atypical Parkinsonism; Dystonia
Keywords: Botulinum toxinum; Dystonia; Parkinson Disease; Atypical Parkinsonism
MeSH Terms: conditions — Parkinson Disease; Dystonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with dystonia secondary to atypical Parkinsonism or Parkinson's disease: Patients with dystonia secondary to idiopathic Parkinson's disease or atypical parkinsonism and treated with BoNT
- Patients with atypical Parkinsonism or Parkinson's disease and no dystonia: Patients with idiopathic Parkinson's disease or atypical parkinsonism and without reported dystonia

SUMMARY:
Dystonia is a disabling symptom affecting both patients with idiopathic Parkinson's disease (PD) and atypical parkinsonism (AP).

Botulinum toxinum (BoNT), by blocking muscle contraction, is a possible treatment for focal dystonia.

The benefit of BoNT treatment has been proven in some focal dystonia associated with PD or AP.

The investigators aim to give an overview of the efficacy of BoNT in a variety of focal dystonia in a large cohort of parkinsonian patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Parkinson's disease or Atypical Parkinsonism
* Age > 18 years
* Reported dystonia
* At least 1 injection with Botulinum toxin realized

Exclusion Criteria:

* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that have been evaluated in the Neurology department of Avicenne Hospital (academic medical center) between september 1st 2017 and february 11th 2021.
  Data will be retrospectively collected within the medical records of those patients.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-02-11 (Actual); Study Completion 2021-02-11 (Actual)

PRIMARY OUTCOMES:
Comparison of the patient reported efficacy of botulinum toxin treatment between PD and AP patients | Up to twelve months
  Evaluation by the patient of the efficacy of the former injection on an improvement scale ranging from 0 to 100% (minimum value : 0, maximum value : 100, higher scores mean a better outcome) systematically made in routine care during follow up appointment

SECONDARY OUTCOMES:
Comparison of the patient reported duration of improvement after treatment by botulinum toxin between PD and AP patients | Up to twelve months
  Evaluation by the patient of the duration of the period during which symptoms were improved (in weeks) systematically made in routine care during follow up appointment

OTHER OUTCOMES:
Comparison of the patients' age between PD and AP groups | Baseline
  Age in years of patients from PD and AP groups
Comparison of the sex-ratio between PD and AP groups | Screening
  Percentage of female (%) in PD and AP groups
Comparison of the patients' duration of disease between PD and AP groups | Baseline
  Duration of the disease (years since diagnosis of PD or AP) of patients from PD and AP groups
Comparison of the patients' severity of the disease between PD and AP groups | Baseline
  Severity of the disease in both PD and AP groups measured by the Hoehn and Yahr scale (stage 0 to stage 5, a higher score meaning a more severe disease)
Comparison of the patients' daily need in levodopa between PD and AP groups | Baseline
  Levodopa equivalent daily dose (in mg, method as described by CL Tomlinson) of patient from PD and AP groups
Comparison of the percentage of patients treated with an apomorphine pump between PD and AP groups | Baseline
  Percentage of patients treated with apomorphine (%) in PD and AP groups
Comparison of the percentage of patients treated with deep brain stimulation between PD and AP groups | Baseline
  Percentage of patients treated with deep brain stimulation (%) in PD and AP groups
Comparison of the patients' age between patients presenting with dystonia and patients without reported dystonia | Baseline
  Age in years
Comparison of the percentage of patients treated with deep brain stimulation between patients presenting with dystonia and patients without reported dystonia | Baseline
  Percentage of patients treated with deep brain stimulation (%) in both groups
Comparison of the percentage of patients treated with an apomorphine pump between patients presenting with dystonia and patients without reported dystonia | Baseline
  Percentage of patients treated with apomorphine (%) in both groups
Comparison of the patients' daily need in levodopa between patients presenting with dystonia and patients without reported dystonia | Baseline
  Levodopa equivalent daily dose (in mg, method as described by CL Tomlinson) of patient from both groups
Comparison of the severity of the disease between patients presenting with dystonia and patients without reported dystonia | Baseline
  Severity of the disease in both groups measured by the Hoehn and Yahr scale (stage 0 to stage 5, a higher score meaning a more severe disease)
Comparison of the patients' duration of disease between patients presenting with dystonia and patients without reported dystonia | Baseline
  Duration of the disease (years since diagnosis of AP or PD) of patients
Comparison of the sex-ratio between patients presenting with dystonia and patients without reported dystonia | Baseline
  Percentage of female (%)
Comparison of the dystonia's characteristics between PD and AP groups : muscle affected | Day 0
  Muscle affected by dystonia (described with International Anatomical Terminology)
Comparison of the dystonia's characteristics between PD and AP groups : duration of dystonia | Day 0
  Duration of the dystonia (years since first report of the dystonia)
Comparison of the characteristics of the botulinum toxin injection between PD and AP groups : dose | Day 0
  Dose of BoNT used (in mL)
Comparison of the characteristics of the botulinum toxin injection between PD and AP groups : type of BoNT | Day 0
  Type of botulinum toxin used (onabotulinumtoxinA, abobotulinumtoxinA or incobotulinumtoxinA)
Comparison of the characteristics of the botulinum toxin injection between PD and AP groups : site of injection | Day 0
  Site of injection (described with International Anatomical Terminology)
Comparison of the characteristics of the botulinum toxin injection between PD and AP groups : number of injections | Day 0
  Number of injection performed during injection appointment
Comparison of the characteristics of the botulinum toxin injection between PD and AP groups : usage of electromyographic or ultrasound guidance | Day 0
  Usage of ultrasound or electromyography to guide BoNT injection

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Degos, MD,PhD, Principal Investigator — Hospital Avicenne
Locations (1):
- Avicenne Hospital, Bobigny, Seine-Saint-Denis, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dressler D. Botulinum toxin drugs: brief history and outlook. J Neural Transm (Vienna). 2016 Mar;123(3):277-9. doi: 10.1007/s00702-015-1478-1. Epub 2015 Nov 11. PMID 26559824
- [Background] Jankovic J. Botulinum toxin: State of the art. Mov Disord. 2017 Aug;32(8):1131-1138. doi: 10.1002/mds.27072. Epub 2017 Jun 22. PMID 28639368
- [Background] Tolosa E, Compta Y. Dystonia in Parkinson's disease. J Neurol. 2006 Dec;253 Suppl 7:VII7-13. doi: 10.1007/s00415-006-7003-6. PMID 17131231
- [Background] Marsili L, Bologna M, Kojovic M, Berardelli A, Espay AJ, Colosimo C. Dystonia in atypical parkinsonian disorders. Parkinsonism Relat Disord. 2019 Sep;66:25-33. doi: 10.1016/j.parkreldis.2019.07.030. Epub 2019 Jul 23. PMID 31443953
- [Background] Mills R, Bahroo L, Pagan F. An update on the use of botulinum toxin therapy in Parkinson's disease. Curr Neurol Neurosci Rep. 2015 Jan;15(1):511. doi: 10.1007/s11910-014-0511-3. PMID 25407133
- [Background] Pacchetti C, Albani G, Martignoni E, Godi L, Alfonsi E, Nappi G. "Off" painful dystonia in Parkinson's disease treated with botulinum toxin. Mov Disord. 1995 May;10(3):333-6. doi: 10.1002/mds.870100317. PMID 7651452
- [Background] Giladi N, Meer J, Honigman S. The use of botulinum toxin to treat "striatal" toes. J Neurol Neurosurg Psychiatry. 1994 May;57(5):659. doi: 10.1136/jnnp.57.5.659. No abstract available. PMID 8201355
- [Background] Rieu I, Degos B, Castelnovo G, Vial C, Durand E, Pereira B, Simonetta-Moreau M, Sangla S, Fluchere F, Guehl D, Burbaud P, Geny C, Gayraud D, Ory-Magne F, Bouhour F, Llinares E, Derost P, Marques A, Durif F. Incobotulinum toxin A in Parkinson's disease with foot dystonia: A double blind randomized trial. Parkinsonism Relat Disord. 2018 Jan;46:9-15. doi: 10.1016/j.parkreldis.2017.10.009. Epub 2017 Oct 19. PMID 29102441
- [Derived] Lapostolle A, Houot M, Mongin M, Degos B. Comparison of Botulinum neurotoxin efficiency in dystonia associated with Parkinson's disease and atypical parkinsonism: a retrospective study with a self-reported improvement scale. J Neurol. 2022 Nov;269(11):6021-6028. doi: 10.1007/s00415-022-11280-y. Epub 2022 Jul 19. PMID 35854137